CLINICAL TRIAL: NCT02378766
Title: Evaluation of a Tailored Virtual Intervention as an Instrument of Prevention and Support to Improve the Health of PLHIV and Reduce Comorbidity Associated With HIV (MP-02-2015-5853)
Brief Title: Evaluation of Web-based Interventions to Support People Living With HIV in the Adoption of Health Behaviors
Acronym: LHIVEHEALTHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CE 14.342
Record Dates: First submitted 2015-02-17; First posted 2015-03-04 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2022-01

CONDITIONS: HIV
Keywords: tailored web-based intervention; health behavior; hiv comorbidities; online trial
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Website A (Experimental): Patients assigned to this arm will be invited to complete a web-based tailored intervention called TAVIE en santé.
  Interventions: Behavioral: Website A
- Website B (Other): Patients assigned to this arm will be invited to consult a validated list of five predetermined websites.
  Interventions: Other: Website B

INTERVENTIONS:
Behavioral: Website A — Patients assigned to this arm will be invited to complete a web-based tailored intervention called TAVIE en santé (TAVIE : Traitement, Assistance Virtuelle Infirmière et Enseignement).
  TAVIE en santé is a web-based tailored multicomponent intervention addressing smoking cessation, physical activity and healthy eating. Each component consists of seven interactive computer sessions lasting 5-10 minutes. The sessions, hosted by a virtual nurse, aims to develop and strengthen skills required for behavior change.
  Arms: Website A
Other: Website B — Patients assigned to this arm will be invited to consult a validated list of five predetermined websites offering information about the health behavior they chose: being physically active, following a healthy diet or quitting smoking. These websites offers reliable information and their content were validated by experts.
  Arms: Website B

SUMMARY:
The purpose of this study is to evaluate the efficacy of a web-based tailored intervention to support persons living with HIV (PLHIV) manage the demands inherent to their health condition, particularly as regards to the adoption of health behaviours such as being physically active, following a healthy diet and quitting smoking.

This randomized controlled trial is currently conducted entirely online at www.lhivehealthy.ca

DETAILED DESCRIPTION:
This online randomized controlled trial with parallel-groups is conducted across Canada. Interested participants are invited to visit the study's Website at www.lhivehealthy.ca

The study's Website contains video clips explaining the study. After accepting the conditions and consenting, participants will enroll in the study by providing an email address and a pseudonym. Each participant will be validated through an email address check. After their enrolment, participants will receive a hyperlink via email to invite them to complete a baseline questionnaire.

After completing the baseline questionnaire, participants will be randomly assigned by the computer system either to an experimental group (TAVIE en santé) or to a control group (list of 5 websites).

Three and six months after the baseline questionnaire, participants will complete the online questionnaires again.

ELIGIBILITY:
Inclusion Criteria:

* to be living with HIV
* to be able to read and understand French or English
* to have access to the Internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Change in tobacco smoking | 6 months
  Measured with a single question: "In the past 7 days, have you had a smoke or even just a single puff? (0=no/1=yes)". Compared to biochemical verification (urinary cotinine test), this self-report measure has a sensitivity of 96.9% and a specificity of 93.4% (Noonan, Jiang et al. 2013) and it correlates well with biochemical validation (Velicer, Prochaska et al. 1992).
Change in level of physical activity | 6 months
  The level of physical activity will be measured through the adaptation of a procedure elaborated and validated by Godin and al. (1985, 1986). Participants will indicate, during a typical week and for each level of intensity (high, moderate, low), the frequency and the mean duration of physical activity practice.
Change in diet quality | 6 months
  Measured with the brief tool Starting The Conversation an 8-item simplified food frequency instrument (Paxton, Strycker et al. 2011) derived from a validated 54-item instrument (Jilcott, Keyserling et al. 2007). Item scores are tallied for an overall score (range of 0-16). STC is stable over time and sensitive to treatment/intervention.

SECONDARY OUTCOMES:
Change in Intention regarding the adoption of the chosen health behaviour | 6 months
  Intention is assessed by three items: 1) "I intend to (a: stop smoking, b: do more physical activity, c: make better choices regarding fat in my diet)" rated on a scale from 1 = strongly disagree to 5 = strongly agree; 2) "I will (a, b or c)" rated on a scale from 1 = very unlikely to 5 = very likely; 3) "the chances that I will (a, b or c) are…" rated on a scale from 1 = very low to 5 = very high. Intention item scores are tallied for an overall score (range of 3-15).
Change in perceived control regarding the adoption of the chosen health behaviour | 6 months
  Perceived control is assessed by three items : 1) "I feel that I will be able to (a: stop smoking, b: do more physical activity, c: make better choices regarding fat in my diet)" rated on a scale from 1 = strongly disagree to 5 = strongly agree; 2) "I am confident that I will succeed in (a, b or c)" rated on a scale from 1 = strongly disagree to 5 = strongly agree; 3) "how much control do you have over (a, b or c)?" rated on a scale from 1 = strongly uncontrollable to 5 = strongly controllable. Perceived control item scores are tallied for an overall score (range of 3-15).
Change in attitude regarding the adoption of the chosen health behaviour | 6 months
  Attitude is measured by asking participants to respond-using five 5-point adjective pairs (unpleasant/pleasant, useless/useful, bad/good, unsatisfying/satisfying, boring/interesting) to the statement linked to their chosen behavior, "Smoking cessation would be for me…" or "Doing more physical activity would be for me…" or "Making better choices regarding fat in my diet would be for me…". Attitude item scores are tallied for an overall score (range of 5-25).

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Cosette, Ph.D., Principal Investigator — Institut de Cardiologie de Montréal; Cécile Tremblay, Md, Ph.D., Principal Investigator — CR-CHUM; Michal Abrahamowicz, Ph.D., Study Chair — McGill University; François Boudreau, Ph.D., Study Chair — Université du Québec à Trois-Rivièves; Jean-Louis Chiasson, Md, Study Chair — CR-CHUM; Alexandra De Pokomandy, Md, Study Chair — CUSM; Marie-Pierre Gagnon, Ph.D., Study Chair — Laval University; Yann-Gaël Guéhéneuc, Ph.D., Study Chair — École Polytechnique de Montréal; Joyal Miranda, Ph.D., Study Chair — Toronto Metropolitan University; Pilar Ramirez-Garcia, Ph.D., Study Chair — Université de Montréal; Catherine Worthington, Ph.D., Study Chair — University of Victoria; José Côté, Ph.D., Principal Investigator — CR-CHUM, Université de Montréal
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Background] Cote J, Cossette S, Ramirez-Garcia P, De Pokomandy A, Worthington C, Gagnon MP, Auger P, Boudreau F, Miranda J, Gueheneuc YG, Tremblay C. Evaluation of a Web-based tailored intervention (TAVIE en sante) to support people living with HIV in the adoption of health promoting behaviours: an online randomized controlled trial protocol. BMC Public Health. 2015 Oct 12;15:1042. doi: 10.1186/s12889-015-2310-4. PMID 26458508